CLINICAL TRIAL: NCT04945889
Title: La Sepsi Nel Paziente Anziano: Studio Prospettico Sui Pazienti Ricoverati in Ambiente Internistico.
Brief Title: Sepsis in Geriatric Patients With Suspected Infection.
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Mario Bo, Director, S.C. Geriatria U, Molinette Hospital, A.O.U. Città della Salute e della Scienza
Other Study IDs: 0069708/2019
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Sepsis
Keywords: Sepsis; Diagnostic accuracy; Geriatric patients; Older adults; Early Warning Score; qSOFA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric inpatients at risk for sepsis: Consecutive patients admitted to an Acute Geriatric Unit for any reason presenting at least one National Institute for Health and Care Excellence (NICE) risk factor for sepsis (age ≥75 years, impaired immune function, long-term corticosteroid therapy, immunosuppressive or antineoplastic drug treatment, surgery or other invasive procedures within 6 weeks, any breach of skin integrity, intravenous drug misuse, indwelling lines or catheters).
  In those with suspected infection (i.e. antibiotic prescription and a culture test within 24 hours before-72 hours after), clinical parameters (respiratory rate, blood pressure, heart rate, body temperature, peripheral oxygen saturation, mental status) were assessed at least twice daily throughout hospital stay and used by study investigators to determine the qSOFA, NEWS and MEWS.
  Interventions: Diagnostic Test: Quick Sequential Organ Failure Assessment (qSOFA); Diagnostic Test: Modified Early Warning Score (MEWS); Diagnostic Test: National Early Warning Score (NEWS)

INTERVENTIONS:
Diagnostic Test: Quick Sequential Organ Failure Assessment (qSOFA) — Clinical bedside tool that evaluates three vital parameters, scoring one point each if altered: respiratory rate (RR) ≥22 breaths/minute, systolic blood pressure (SBP) ≤100 mmHg and altered mental status (defined in our study as either Glasgow Coma Scale (GCS) score <15 or any worsening in the Italian Oriented, Disoriented, Agitated, Sleepy scale). A qSOFA score ≥2 points is considered indicative of sepsis.
  Other Names: Quick Sepsis-Related Organ Failure Assessment
Diagnostic Test: Modified Early Warning Score (MEWS) — Clinical bedside tool that evaluates five vital parameters, with multiple scoring according to alteration: respiratory rate (0-3 points), heart rate (0-3 points), systolic blood pressure (0-3 points), body temperature (0-2 points), mental status (0-3 points, evaluated using the Alert, Verbal, Pain, Unresponsive - AVPU scale). A MEWS score ≥5 points is considered indicative of an acute condition at risk of sudden clinical deterioration.
Diagnostic Test: National Early Warning Score (NEWS) — Clinical bedside tool that evaluates seven parameters, with multiple scoring according to alteration: respiratory rate (0-3 points), oxygen saturation (0-3 points), need for any supplemental oxygen (0-2 points), body temperature (0-3 points), heart rate (0-3 points), systolic blood pressure (0-3 points), mental status (0-3 points, evaluated using the Alert, Verbal, Pain, Unresponsive - AVPU scale). A NEWS score ≥7 points is considered indicative of an acute condition at risk of sudden clinical deterioration.

SUMMARY:
Sepsis is a complex clinical syndrome that has been defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection. It is more frequent and severe in older subjects, at least in part because of delayed diagnosis and treatment due to low clinical suspicion and atypical manifestation.

The Sepsis-III consensus proposed the easy to use bedside clinical score quick Sequential Organ Failure Assessment (qSOFA) to identify patients at risk for sepsis and death outside intensive care units. However, some Authors have disputed this recommendation, proposting the use of other more complex bedside tools such as the National and Modified Early Warning Scores (NEWS and MEWS, respectively) for the same purpose.

Published studies on these scores included generally younger, selected subjects, not fully representative of the population at risk for sepsis.

In the present study we aimed to evaluate the incidence of sepsis in older subjects with suspected infection in a geriatric acute ward setting, to determine and compare the accuracies of qSOFA, NEWS and MEWS to identify sepsis and to investigate factors associated with in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the Acute Geriatric Unit
* Presence of at least one National Institute for Health and Care Excellence (NICE) guidance risk factor for sepsis (i.e. age ≥75 years, impaired immune function - diabetes mellitus, previous splenectomy, hematologic diseases - long-term corticosteroid therapy, immunosuppressive or antineoplastic drug treatment, surgery or other invasive procedures in the previous 6 weeks, any breach of skin integrity - e.g. pressure ulcers - intravenous drug misuse, indwelling lines or catheters)

Exclusion Criteria:

* Refusal to give written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients admitted for any cause, to an acute geriatric ward of a large university teaching hospital in North-western Italy, with at least one NICE risk factor for sepsis, providing written informed consent. Intervention (diagnostic test administration) was performed only in patients with a suspected infection, defined as the prescription of an oral and/or parenteral antibiotic therapy within a timeframe spanning from 24 hours before and 72 hours after the collection of a biological sample to perform a culture test.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Sepsis diagnosis at discharge | 10 days from enrollment in mean (discharge from hospital)
  Presence in discharge documents of International Classification of Diseases 9th revision, Clinical Modification (ICD-9-CM) codes at discharge of either severe sepsis (995.92) or septic shock (785.52) or as the simultaneous presence in discharge documents of ICD-9-CM codes of infection and at least one acute organ dysfunction (Angus method).

OTHER OUTCOMES:
In hospital mortality | 10 days from enrollment in mean (discharge from hospital)
  Presence in discharge documents of death during hospital stay for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bo, MD, PhD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- S.C. Geriatria U, A.O.U. Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Result] Rowe TA, McKoy JM. Sepsis in Older Adults. Infect Dis Clin North Am. 2017 Dec;31(4):731-742. doi: 10.1016/j.idc.2017.07.010. PMID 29079157
- [Result] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Result] Song JU, Sin CK, Park HK, Shim SR, Lee J. Performance of the quick Sequential (sepsis-related) Organ Failure Assessment score as a prognostic tool in infected patients outside the intensive care unit: a systematic review and meta-analysis. Crit Care. 2018 Feb 6;22(1):28. doi: 10.1186/s13054-018-1952-x. PMID 29409518
- [Result] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Result] Smith GB, Prytherch DR, Meredith P, Schmidt PE, Featherstone PI. The ability of the National Early Warning Score (NEWS) to discriminate patients at risk of early cardiac arrest, unanticipated intensive care unit admission, and death. Resuscitation. 2013 Apr;84(4):465-70. doi: 10.1016/j.resuscitation.2012.12.016. Epub 2013 Jan 4. PMID 23295778
- [Result] Kramer AA, Sebat F, Lissauer M. A review of early warning systems for prompt detection of patients at risk for clinical decline. J Trauma Acute Care Surg. 2019 Jul;87(1S Suppl 1):S67-S73. doi: 10.1097/TA.0000000000002197. PMID 31246909
- See also: NICE sepsis guidance — https://www.nice.org.uk/guidance/ng51
- See also: NEWS — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&ved=2ahUKEwia9qjN-LnxAhXFzaQKHfyrAL8QFjABegQIAhAD&url=https%3A%2F%2Fwww.rcplondon.ac.uk%2Ffile%2F32%2Fdownload%3Ftoken%3D5NwjEyTq&usg=AOvVaw1pY4NhC88X7yoJziKB3odI